CLINICAL TRIAL: NCT07116759
Title: Real-Time Head Position Stabilization of Healthy Volunteers
Brief Title: Head Stabilization of Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UPCC 07325; R01CA227124-02 (NIH); 843058 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2025-08-07; First posted 2025-08-12 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy Volunteers: The volunteer population will consist of healthy individuals.
  Interventions: Device: Real-time head stabilization with robotic platform

INTERVENTIONS:
Device: Real-time head stabilization with robotic platform — A robotic platform will use data from motion-detection cameras to position a person's head in real time. This procedure is non-invasive.

SUMMARY:
A robotic platform will use data from motion-detection cameras to position a person's head in real time. This procedure is non-invasive and since healthy volunteers are enrolled in this study, no radiation is delivered, but in the future, the investigators plan to use this device during radiation treatment with patients.

DETAILED DESCRIPTION:
This study aims to passively monitor the real-time head motions of healthy volunteers positioned to simulate whole brain radiation therapy. Such real-time head motion data is necessary in order to understand the type (amplitude/frequency) of motion that the robotic stage will be expected to compensate for and will play an important role in the overall modeling and designing process of the robotic prototype.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 and older
* Subjects must be able to read and understand English
* Participants must sign the informed consent form

Exclusion Criteria:

Any subjects not meeting the above inclusion criteria will not be considered for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The volunteer population will consist of healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-10-09 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Wiersma, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 20
Completed | 18
Not Completed | 2
Not completed — Incompatibility with the RHMC device | 2

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Collection of Head Motion Data to be Used in Developing Head Stabilization Methods in Brain Radiation Patients
Description: Real-time intracranial target motion was continuously monitored using a commercial surface-guided radiation therapy (SGRT) system operating at approximately 10 frames per second. For each participant, translational (mm) and rotational (degree) motion of the target were computed relative to the starting head position at setup. The target position was tracked in six degrees of freedom (longitudinal, lateral, vertical translation; pitch, roll, yaw rotation). To provide a quantitative endpoint reflecting system effectiveness, the recorded 6D target motion data were analyzed and positional deviation histograms showing the total percentage of time that the target remained below a specific translational and rotational tolerance level were generated. The percentage of time that the target remained below a tolerance of < 1.0 mm translational and < 1.0° rotational deviation was chosen as the single primary outcome measure.
Time Frame: One-time session, up to 4 hours on a single day.
Population: 18 healthy volunteers, who successfully completed simulating in a clinical environment but without delivering radiation
Measure: Mean (95% Confidence Interval); unit: % of time within tolerance
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 18
% of time within tolerance | 95 [80 to 100]

ADVERSE EVENTS:
Time Frame: 1 year and 6 months
Arm/Group | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT07116759/Prot_SAP_000.pdf